CLINICAL TRIAL: NCT01866501
Title: A Follow-up Study Validating a Blended Technique for Identifying the Proximal Humerus Intraosseous Vascular Access Insertion Site
Brief Title: Follow-Up Study Validating a Blended Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vidacare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2013-06
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Intraosseous Vascular Access
Keywords: Intraosseous Vascular Access; IO Access; IO Vascular Access; EZ-IO
MeSH Terms: interventions — Jupiter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blended Technique (Experimental): Using the blended technique device operators will establish proximal humerus intraosseous vascular access.
  Interventions: Procedure: Proximal Humerus Intraosseous Vascular Access; Device: EZ-IO

INTERVENTIONS:
Procedure: Proximal Humerus Intraosseous Vascular Access — Using the blended technique, device operators will establish proximal humerus intraosseous vascular access by inserting an IO needle.
  Other Names: EZ-IO; Intraosseous Vascular Access; Proximal Humerus IO Access; IO
Device: EZ-IO

SUMMARY:
A Follow-up Study Validating a Blended Technique for Identifying the Proximal Humerus Intraosseous Vascular Access Insertion Site

DETAILED DESCRIPTION:
In 2012, the investigators from Vidacare evaluated 4 techniques commonly used to identify the proximal humerus IO insertion site to determine if one technique resulted in more consistent successful placement of the IO needle set with a higher level of confidence among device operators performing the techniques. Results suggest that a combination of the best features of the 4 techniques may lead to optimal IO needle set placement more consistently. This study is needed to validate the "Blended" proximal humerus IO insertion technique to confirm that use of the technique results in proper site identification among device operators and results in increased confidence.To most closely evaluate the Blended proximal humerus insertion technique and how it is received by clinicians who perform these procedures in actual patients, device operators will include licensed/certified clinicians including, emergency medicine technicians/paramedics and nurses.

ELIGIBILITY:
Inclusion Criteria:

* Currently licensed/certified Emergency Medicine Technicians, paramedic, or nurse Have had no formal training on use of the proximal humerus IO insertion site Demonstrate proper use of the device and technique during training portion and obtain approval from the device trainer to participate

Exclusion Criteria:

* Previous training on establishing proximal humerus intraosseous vascular access

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Successful IO insertion | Day 1 after establishing proximal humerus IO vascular access
  Successful IO needle insertion determined by x-ray images

SECONDARY OUTCOMES:
Intraosseous Infusion flow rates | Day 1 after establishing IO vascular access
  Intraosseous infusion flow rates attained using 4 different infusion pressures Gravity; 100 mmHg, 200 mmHg and 300 mmHg.
Time in seconds for fluid delivery from the proximal humerus to the heart, using visualization of contrast injection under fluoroscopy. | Day 1 after IO insertion
Relationship between IO and peripheral venous blood | Day 1 after establishing IO vascular access and peripheral venous access
  IO blood and peripheral venous blood will be collected and analyzed for routine blood tests and the results will be compared to determine if there is a relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Larry J Miller, MD, Principal Investigator — Vidacare Corporation
Locations (1):
- Bulverde-Spring Branch EMS, Spring Branch, Texas, United States